CLINICAL TRIAL: NCT04024436
Title: A Phase 2 Study of TAS-120 in Metastatic Breast Cancers Harboring Fibroblast Growth Factor Receptor (FGFR) Amplifications
Brief Title: A Study of TAS-120 in Patients With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor decided to discontinue the study due to strategic considerations and not due to any safety-related concerns.
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FOENIX-MBC2 TAS-120-201; 2019-001164-30 (EudraCT Number)
Record Dates: First submitted 2019-06-24; First posted 2019-07-18 (Actual); Results first posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Breast Cancer; FGFR 1 High Amplification; FGFR2 Amplification
Keywords: Futibatinib; Metastatic Breast Cancer; FGFR; TAS-120
MeSH Terms: conditions — Breast Neoplasms | interventions — futibatinib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Futibatinib (Cohort 1) (Experimental): Participants with advanced or metastatic hormone receptor - positive (HR+), human epidermal growth factor receptor 2 - negative (HER2-) breast cancer, harboring fibroblast growth factor receptor 2 (FGFR2) gene amplification, with measurable disease received futibatinib, 20 milligrams (mg), oral tablets, once daily for a continuous 28-day cycle up to maximum of 244 days.
  Interventions: Drug: Futibatinib
- Futibatinib (Cohort 2) (Experimental): Participants with advanced or metastatic triple negative breast cancer (TNBC), harboring FGFR2 gene amplification, with measurable disease received futibatinib, 20 mg, oral tablets, once daily for a continuous 28-day cycle up to maximum of 1066 days.
  Interventions: Drug: Futibatinib
- Futibatinib (Cohort 3) (Experimental): Participants with advanced or metastatic HR+, HER2- or TNBC, harboring FGFR2 gene amplification, with non-measurable disease received futibatinib, 20 mg, oral tablets, once daily for a continuous 28-day cycle up to maximum of 252 days.
  Interventions: Drug: Futibatinib
- Futibatinib Plus Fulvestrant (Cohort 4) (Experimental): Participants with advanced or metastatic HR+ HER2- breast cancer, harboring FGFR1 gene amplification, with measurable disease, received futibatinib, 20 mg, oral tablets, once daily for a continuous 28-day cycle up to maximum of 645 days. They also received intramuscular (IM) fulvestrant 500 mg on Days 1 and 15 of Cycle 1 and Day 1 of every subsequent cycle up to maximum of 618 days.
  Interventions: Drug: Futibatinib plus Fulvestrant

INTERVENTIONS:
Drug: Futibatinib — Futibatinib 20mg once daily on a 28-day cycle
  Other Names: TAS-120
  Arms: Futibatinib (Cohort 1); Futibatinib (Cohort 2); Futibatinib (Cohort 3)
Drug: Futibatinib plus Fulvestrant — Futibatinib 20mg once daily on a 28-day cycle and fulvestrant 500 mg administered intramuscularly (IM) on Days 1 and 15 of Cycle 1, then on Day 1 of Cycle 2 and beyond on a 28-day cycle.
  Arms: Futibatinib Plus Fulvestrant (Cohort 4)

SUMMARY:
The purpose of the trial is to evaluate a patient's response to a Fibroblast Growth Factor Receptor (FGFR) inhibitor, futibatinib (TAS-120), used either alone or in combination with the hormonal therapy, fulvestrant. This study will be conducted in patients with metastatic breast cancer who have specific Fibroblast Growth Factor Receptor gene abnormalities and who have previously received conventional therapies to treat their breast cancer, or who are not able to tolerate certain cancer therapies. This study will also evaluate the safety of taking futibatinib, or futibatinib and fulvestrant, by learning about the potential side effects.

DETAILED DESCRIPTION:
This is a Phase 2, open-label, non-randomized, multicenter study designed to evaluate the efficacy and safety of futibatinib (TAS-120) and futibatinib + fulvestrant in up to 168 adult patients with locally advanced/metastatic breast cancer harboring FGFR gene amplifications. Patients will be enrolled to 1 of 4 treatment cohorts based on diagnosis and FGFR gene amplification status, and will receive either single agent futibatinib in Cohorts 1-3 or futibatinib plus fulvestrant in Cohort 4, as follows:

* Cohort 1 - HR+ HER2- Measurable Disease w/ FGFR2 Amplification
* Cohort 2 - TNBC Measurable Disease w/ FGFR2 Amplification
* Cohort 3 - HR+ HER2- or TNBC Non-Measurable Disease w/ FGFR2 Amplification
* Cohort 4 - HR+ HER2- Measurable Disease w/ FGFR1 Amplification

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. Age ≥ 18 years of age
3. Histologically or cytologically confirmed recurrent locally advanced or metastatic breast cancer not amenable to treatment with curative intent, and the following cohort specific criteria:

   A. Cohort 1
   * HR+ HER2- breast cancer harboring an FGFR2 gene amplification.
   * Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
   * Has received 1-3 prior endocrine-containing therapies and up to 2 prior chemotherapy regimens for advanced/metastatic disease
   * Has received prior treatment with a CDK4/6 inhibitor or is ineligible for such treatment

   B. Cohort 2
   * TNBC harboring an FGFR2 gene amplification
   * Measurable disease per RECIST 1.1
   * Has received at least 1 prior chemotherapy or chemotherapy/immunotherapy (PD-L1/PD-1 inhibitors) regimen for advanced/metastatic disease

   C. Cohort 3
   * TNBC or HR+ HER2- breast cancer harboring an FGFR2 gene amplification
   * Non measurable, evaluable disease per RECIST 1.1. Patients with bone-only disease must have lytic or mixed lytic-blastic lesions
   * Other criteria for either HR+ HER2- breast cancer or TNBC should be met as described for Cohort 1 and 2, respectively

   D. Cohort 4
   * HR+ HER2- breast cancer harboring an FGFR1 high-level gene amplification
   * Measurable disease per RECIST 1.1
   * Has received 1-2 prior endocrine-containing therapies and no more than 1 prior chemotherapy regimen for advanced/metastatic disease. Prior treatment with fulvestrant is not permitted.
   * Has received prior treatment with a CDK4/6 inhibitor or is ineligible for such treatment
   * Pre/peri-menopausal patients must be on goserelin
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
5. Archival or (preferably) fresh tumor tissue must be available
6. Adequate organ function

Exclusion Criteria:

1. History and/or current evidence of any of the following disorders:

   1. Non-tumor related alteration of the calcium-phosphorus homeostasis that is considered clinically significant
   2. Ectopic mineralization/calcification, including but not limited to soft tissue, kidneys, intestine, or myocardia and lung, considered clinically significant
   3. Retinal or corneal disorder confirmed by retinal/corneal examination and considered clinically significant
2. Prior treatment with an FGFR inhibitor
3. A serious illness or medical condition(s)
4. Brain metastases that are untreated or clinically or radiologically unstable
5. Pregnant or lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-09-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (17):
  - Mayo Clinic - AZ, Phoenix, Arizona
  - USCF, San Francisco, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Mayo Clinic - FL, Jacksonville, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Florida Cancer Specialists, Tallahassee, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - BIDMC, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic - MN, Rochester, Minnesota
  - HCA Midwest Health, Kansas City, Missouri
  - Tennessee Oncology, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - MD Anderson, Houston, Texas
- Canada (2):
  - Tom Baker Cancer Center, Calgary
  - SunnyBrook Health Sciences, Toronto
- France (2):
  - Institut Gustave Roussy, Villejuif, Cedex
  - Centre Leon Berard, Lyon
- Italy (7):
  - AOU Policlinico - Vittorio Emanuele, Catania
  - Istituto Europeo Di Oncologia - IEO, Milan
  - AOU Modena Policlinico, Modena
  - Ospedale E. Agnelli, Pinerolo
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Portugal (3):
  - Centro Hospitalar Universitario Lisboa Norte, Lisbon
  - Porto University, Porto
  - Instituto Portugues de Oncologia do Porto, Porto
- Spain (3):
  - Vall d'Hebron, Barcelona
  - University Gregorio Marañon, Madrid
  - START Madrid - CIOCC, Madrid
- United Kingdom (3):
  - HCA Healthcare UK, London, England
  - The Christie NHS Foundation Trust, Manchester, England
  - The Royal Marsden NHS Foundation Trust, Sutton, England

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study from 28 January 2020 to 06 September 2023.
Pre-assignment Details: A total of 64 participants were enrolled in either Cohorts 1, 2 or 3 to receive futibatinib or to Cohort 4 to receive futibatinib plus fulvestrant.
Groups:
- Futibatinib Plus Fulvestrant (Cohort 4): Participants with advanced or metastatic HR+ HER2- breast cancer, harboring FGFR1 gene amplification, with measurable disease, received futibatinib, 20 mg, oral tablets, once daily for a continuous 28-day cycle up to maximum of 645 days. They also received IM fulvestrant 500 mg on Days 1 and 15 of Cycle 1 and Day 1 of every subsequent cycle up to maximum of 618 days.
Period: Overall Study
Arm/Group | Futibatinib (Cohort 1) | Futibatinib (Cohort 2) | Futibatinib (Cohort 3) | Futibatinib Plus Fulvestrant (Cohort 4)
Started | 17 | 21 | 4 | 22
Completed | 0 | 0 | 0 | 0
Not Completed | 17 | 21 | 4 | 22
Not completed — Death | 10 | 14 | 2 | 7
Not completed — Loss to follow up | 1 | 0 | 0 | 1
Not completed — Withdrawal of consent | 2 | 0 | 0 | 1
Not completed — Study termination by sponsor | 4 | 6 | 2 | 11
Not completed — Reason Not Specified | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All treated population included all enrolled participants who received at least 1 dose of study drug.
Groups:
- Futibatinib (Cohort 1): Participants with advanced or metastatic HR+, HER2- breast cancer, harboring FGFR2 gene amplification, with measurable disease received futibatinib, 20 mg, oral tablets, once daily for a continuous 28-day cycle up to maximum of 244 days
- Futibatinib (Cohort 2): Participants with advanced or metastatic TNBC, harboring FGFR2 gene amplification, with measurable disease received futibatinib, 20 mg, oral tablets, once daily for a continuous 28-day cycle up to maximum of 1066 days.
- Total: Total of all reporting groups
Arm/Group | Futibatinib (Cohort 1) | Futibatinib (Cohort 2) | Futibatinib (Cohort 3) | Futibatinib Plus Fulvestrant (Cohort 4) | Total
Number analyzed (Participants) | 17 | 21 | 4 | 22 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (11.42) | 51.4 (14.50) | 60.8 (5.74) | 52.7 (12.68) | 54.7 (13.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 4 | 22 | 64
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2 | 4
  Not Hispanic or Latino | 15 | 15 | 4 | 13 | 47
  Unknown or Not Reported | 1 | 5 | 0 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 2 | 1 | 0 | 1 | 4
  White | 14 | 12 | 4 | 16 | 46
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 7 | 0 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) - Cohorts 1, 2
Description: ORR was defined as the percentage of participants with a confirmed response of either complete response (CR) or partial response (PR), based on Investigator assessment. CR was defined as disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to <10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of the target lesions, taking as a reference the baseline sum diameters. ORR was calculated based on the best overall response recorded from the start of treatment until progressive disease or start of subsequent new anticancer treatment. Percentages were rounded off to the nearest single decimal place.
Time Frame: At the end of every 2 cycles until disease progression (up to 40 months)
Population: All treated population included all enrolled participants who received at least 1 dose of study drug. This outcome measure was planned to be reported for only Cohort 1 and 2 as pre-specified in Protocol and SAP.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Futibatinib (Cohort 1) | Futibatinib (Cohort 2)
Number analyzed (Participants) | 17 | 21
percentage of participants | 0 [0.0 to 19.5] | 9.5 [1.2 to 30.4]

2. Primary Outcome: Clinical Benefit Rate (CBR) - Cohort 3
Description: CBR was defined as the percentage of participants with a confirmed response of CR or stable disease (SD) lasting at least 24 weeks, based on Investigator assessment. CR was defined as disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to <10mm. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), referencing the smallest sum diameters while on study. PR was defined as at least a 30% decrease in the sum of diameters of the target lesions, taking as a reference the baseline sum diameters. PD was defined as at least a 20% increase in the sum of diameters of the target lesions, taking as a reference the smallest sum on study, including the baseline sum. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Definitive new lesion presence also indicates progression. Percentages were rounded off to the nearest
Time Frame: At the end of every 2 cycles until disease progression (up to 40 months)
Population: All treated population included all enrolled participants who received at least 1 dose of study drug. This outcome measure was planned to be reported for only Cohort 3 as pre-specified in Protocol and SAP.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Futibatinib (Cohort 3)
Number analyzed (Participants) | 4
percentage of participants | 50.0 [6.8 to 93.2]

3. Primary Outcome: 6-month Progression-free Survival (PFS) Rate - Cohort 4
Description: The 6-month PFS rate was defined as the percentage of participants who are alive and progression-free 6 months after the first dose of study drug. Percentages were rounded off to the nearest single decimal place.
Time Frame: At the end of every 2 cycles until disease progression (up to 6 months)
Population: All treated population included all enrolled participants who received at least 1 dose of study drug. This outcome measure was planned to be reported for only Cohort 4 as pre-specified in Protocol and SAP.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Futibatinib Plus Fulvestrant (Cohort 4)
Number analyzed (Participants) | 22
percentage of participants | 45.5 [24.4 to 67.8]

4. Secondary Outcome: Complete Response (CR) Rate - Cohort 3
Description: CR rate was defined as the percentage of participants who achieved CR. CR was defined as disappearance of all targets. Any pathological lymph node must have reduction in short axis to <10 mm. Percentages were rounded off to the nearest single decimal place.
Time Frame: At the end of every 2 cycles until disease progression (up to 40 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Futibatinib (Cohort 3)
Number analyzed (Participants) | 4
percentage of participants | 0 [0.0 to 60.2]

5. Secondary Outcome: Overall Response Rate (ORR) - Cohort 4
Description: ORR was defined as the percentage of participants with a confirmed response of either CR or PR, based on Investigator assessment. CR was defined as disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of the target lesions, taking as a reference the baseline sum diameters. ORR was calculated based on the best overall response recorded from the start of treatment until progressive disease or start of subsequent new anticancer treatment. Percentages were rounded off to the nearest single decimal place.
Time Frame: At the end of every 2 cycles until disease progression (up to 40 months)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Futibatinib Plus Fulvestrant (Cohort 4): Participants with advanced or metastatic HR+ HER2- harboring FGFR1 gene amplification, with measurable disease, received futibatinib, 20 mg, oral tablets, once daily for a continuous 28-day cycle up to maximum of 645 days. They also received IM fulvestrant 500 mg on Days 1 and 15 of Cycle 1 and Day 1 of every subsequent cycle up to maximum of 618 days.
Arm/Group | Futibatinib Plus Fulvestrant (Cohort 4)
Number analyzed (Participants) | 22
percentage of participants | 18.2 [5.2 to 40.3]

6. Secondary Outcome: Clinical Benefit Rate (CBR) - Cohort 1,2, and 4
Description: CBR was defined as the percentage of participants with a confirmed response of CR, PR or SD lasting at least 24 weeks, based on Investigator assessment. CR was defined as disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of the target lesions, taking as a reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, referencing the smallest sum diameters while on study. PD was defined as at least a 20% increase in the sum of diameters of the target lesions, taking as a reference the smallest sum on study, including the baseline sum. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Definitive new lesion presence also indicates progression. Percentages were rounded off to the nearest single decimal place.
Time Frame: At the end of every 2 cycles until disease progression (up to 40 months)
Population: All treated population included all enrolled participants who received at least 1 dose of study drug. This outcome measure was planned to be reported for only Cohorts 1, 2 and 4 as pre-specified in Protocol and SAP.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Futibatinib (Cohort 1) | Futibatinib (Cohort 2) | Futibatinib Plus Fulvestrant (Cohort 4)
Number analyzed (Participants) | 17 | 21 | 22
percentage of participants | 11.8 [1.5 to 36.4] | 23.8 [8.2 to 47.2] | 50.0 [28.2 to 71.8]

7. Secondary Outcome: 6-month PFS Rate - Cohorts 1,2, and 3
Description: as for outcome 3
Time Frame: At the end of every 2 cycles until disease progression (up to 6 months)
Population: All treated population included all enrolled participants who received at least 1 dose of study drug. This outcome measure was planned to be reported for only Cohorts 1, 2 and 3 as pre-specified in Protocol and SAP.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Futibatinib (Cohort 1): Participants with advanced or metastatic HR+, HER2- measurable breast cancer, harboring FGFR2 gene amplification, with measurable disease received futibatinib, 20 mg, oral tablets, once daily for a continuous 28-day cycle up to maximum of 244 days.
- Futibatinib (Cohort 2): Participants with advanced or metastatic TNBC, measurable harboring FGFR2 gene amplification, with measurable disease received futibatinib, 20 mg, oral tablets, once daily for a continuous 28-day cycle up to maximum of 1066 days.
Arm/Group | Futibatinib (Cohort 1) | Futibatinib (Cohort 2) | Futibatinib (Cohort 3)
Number analyzed (Participants) | 17 | 21 | 4
percentage of participants | 5.9 [0.1 to 28.7] | 19.0 [5.4 to 41.9] | 50.0 [6.8 to 93.2]

8. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the first dose of study therapy to the date of death (any cause) or disease progression based on investigator assessment, whichever occurs first. The PFS was analyzed using a Kaplan-Meier method with PFS time being censored on the date of the last disease assessment. The 95% CI for median PFS was provided using the Kaplan-Meier procedure.
Time Frame: At the end of every 2 cycles until disease progression (up to 40 months)
Population: All treated population included all enrolled participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Futibatinib Plus Fulvestrant (Cohort 4): Participants with advanced or metastatic HR+ HER2- breast cancer, harboring FGFR1 gene amplification, with measurable disease, received futibatinib, 20 mg, oral tablets, once daily for a continuous 28-day cycle up to maximum of 645 days.They also received IM fulvestrant 500 mg on Days 1 and 15 of Cycle 1 and Day 1 of every subsequent cycle up to maximum of 618 days.
Arm/Group | Futibatinib (Cohort 1) | Futibatinib (Cohort 2) | Futibatinib (Cohort 3) | Futibatinib Plus Fulvestrant (Cohort 4)
Number analyzed (Participants) | 17 | 21 | 4 | 22
months | 3.7 [1.7 to 5.1] | 1.9 [1.6 to 4.0] | 12.4 [1.9 to NA] — Upper limit of 95% CI was not estimable due to a lack of sufficient number of events within the cohort to estimate the parameter. | 7.2 [2.1 to 7.6]

9. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first documentation of objective response to the to the date of death (any cause) or disease progression, based on Investigator assessment, whichever occurs first. Objective response was defined as participants with a confirmed response of either CR or PR, based on Investigator assessment. CR was defined as disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of the target lesions, taking as a reference the baseline sum diameters. DOR was estimated using the Kaplan-Meier method.
Time Frame: At the end of every 2 cycles until disease progression (up to 40 months)
Population: All treated population included all enrolled participants who received at least 1 dose of study drug. Overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Futibatinib (Cohort 1) | Futibatinib (Cohort 2) | Futibatinib (Cohort 3) | Futibatinib Plus Fulvestrant (Cohort 4)
Number analyzed (Participants) | 0 | 2 | 0 | 4
months |  | 3.38 [3.1 to 3.7] |  | 6.34 [3.3 to 16.7]

10. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time (in months) from the date of first dose of the study drug to the date of death. Participants without a documented death date were censored on the last date they were known to be alive. The OS was presented using a Kaplan-Meier estimate. The 95% CI for median OS was provided using the Kaplan-Meier procedure.
Time Frame: Up to 40 months
Population: All treated population included all enrolled participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Futibatinib (Cohort 1) | Futibatinib (Cohort 2) | Futibatinib (Cohort 3) | Futibatinib Plus Fulvestrant (Cohort 4)
Number analyzed (Participants) | 17 | 21 | 4 | 22
months | 16.5 [8.1 to NA] — Upper limit of 95% CI was not estimable due to a lack of sufficient number of events within the cohort to estimate the parameter. | 10.2 [6.1 to 21.8] | 30.4 [12.4 to NA] — Upper limit of 95% CI was not estimable due to a lack of sufficient number of events within the cohort to estimate the parameter. | 23.9 [20.6 to NA] — Upper limit of 95% CI was not estimable due to a lack of sufficient number of events within the cohort to estimate the parameter.

11. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a clinical study participant and does not necessarily have a causal relationship with the study drug.
Time Frame: From the first dose of study drug up to 30 days after the last dose (Up to 40 months)
Population: All treated population included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Futibatinib (Cohort 2): Participants with advanced or metastatic triple negative breast cancer (TNBC) measurable harboring FGFR2 gene amplification received Futibatinib, 20 mg, oral tablets once daily for a continuous 28-day cycle up to maximum of 1066 days.
Arm/Group | Futibatinib (Cohort 1) | Futibatinib (Cohort 2) | Futibatinib (Cohort 3) | Futibatinib Plus Fulvestrant (Cohort 4)
Number analyzed (Participants) | 17 | 21 | 4 | 22
Participants | 17 | 21 | 4 | 22

12. Secondary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) - Cohort 4
Description: A DLT was defined as any AE that occurs during Cycle 1 that is not clearly attributable to an extraneous cause, such as an underlying disease, occurring in Cycle 1, and meeting at least one of the criteria defined in the protocol. An AE is defined as any untoward medical occurrence in a clinical study participant and does not necessarily have a causal relationship with the study drug.
Time Frame: Cycle 1 (cycle length= 28 days)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Futibatinib Plus Fulvestrant (Cohort 4)
Number analyzed (Participants) | 22
Participants | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 30 days after the last dose (Up to 40 months)
Description: All treated population included all enrolled participants who received at least 1 dose of study drug.
Groups:
- Futibatinib Plus Fulvestrant (Cohort 4): Participants with advanced or metastatic HR+ HER2-, harboring FGFR1 gene amplification, with measurable disease, received futibatinib, 20 mg, oral tablets, once daily for a continuous 28-day cycle up to maximum of 645 days. They also received intramuscular (IM) fulvestrant 500 mg on Days 1 and 15 of Cycle 1 and Day 1 of every subsequent cycle up to maximum of 618 days.
Arm/Group | Futibatinib (Cohort 1) | Futibatinib (Cohort 2) | Futibatinib (Cohort 3) | Futibatinib Plus Fulvestrant (Cohort 4)
All-Cause Mortality (participants affected / at risk) | 10/17 | 14/21 | 2/4 | 7/22
Serious Adverse Events (participants affected / at risk) | 4/17 | 5/21 | 1/4 | 4/22
Other Adverse Events (participants affected / at risk) | 16/17 | 21/21 | 4/4 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Futibatinib (Cohort 1) (N=17) | Futibatinib (Cohort 2) (N=21) | Futibatinib (Cohort 3) (N=4) | Futibatinib Plus Fulvestrant (Cohort 4) (N=22)
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0
Hepatic ischaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Futibatinib (Cohort 1) (N=17) | Futibatinib (Cohort 2) (N=21) | Futibatinib (Cohort 3) (N=4) | Futibatinib Plus Fulvestrant (Cohort 4) (N=22)
Hyperphosphataemia (Metabolism and nutrition disorders) | 13 | 18 | 3 | 21
Decreased appetite (Metabolism and nutrition disorders) | 2 | 4 | 1 | 7
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 3 | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 8 | 9 | 1 | 13
Diarrhoea (Gastrointestinal disorders) | 4 | 8 | 1 | 10
Nausea (Gastrointestinal disorders) | 7 | 6 | 0 | 9
Dry mouth (Gastrointestinal disorders) | 5 | 4 | 1 | 10
Vomiting (Gastrointestinal disorders) | 2 | 4 | 1 | 7
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 1 | 4
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 7 | 5 | 0 | 11
Alanine aminotransferase increased (Investigations) | 4 | 2 | 0 | 13
Weight decreased (Investigations) | 4 | 4 | 1 | 6
Blood alkaline phosphatase increased (Investigations) | 2 | 3 | 1 | 6
Blood bilirubin increased (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 2
White blood cell count decreased (Investigations) | 1 | 1 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 2 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 2 | 0 | 0
Blood phosphorus increased (Investigations) | 1 | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0 | 0
Computerised tomogram abnormal (Investigations) | 1 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 3 | 1 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 6 | 0 | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 5
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 3
Nail discolouration (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 3 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 2 | 5
Headache (Nervous system disorders) | 4 | 2 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 3
Taste disorder (Nervous system disorders) | 1 | 1 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1
Seizure (Nervous system disorders) | 1 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 1
Tremor (Nervous system disorders) | 0 | 1 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 7 | 3 | 7
Asthenia (General disorders) | 0 | 3 | 0 | 3
Mucosal inflammation (General disorders) | 0 | 3 | 0 | 0
Malaise (General disorders) | 0 | 2 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 0 | 0
Dry eye (Eye disorders) | 2 | 5 | 2 | 7
Ocular hyperaemia (Eye disorders) | 1 | 1 | 0 | 1
Vision blurred (Eye disorders) | 1 | 1 | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 1 | 1 | 0 | 0
Central serous chorioretinopathy (Eye disorders) | 1 | 0 | 0 | 0
Corneal disorder (Eye disorders) | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0
Growth of eyelashes (Eye disorders) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 5 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 2
Eye infection (Infections and infestations) | 0 | 2 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 2
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Herpes simplex reactivation (Infections and infestations) | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Oropharyngeal pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The Sponsor decided to discontinue the study due to strategic considerations and not due to any safety-related concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT04024436/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT04024436/SAP_001.pdf